CLINICAL TRIAL: NCT00669617
Title: A Phase III, Randomized, Double-blind, Triple-dummy, Placebo Controlled, Multicenter, 5-period, Single-dose Complete Block Crossover Study to Determine the Onset of Action of Indacaterol (150 and 300 μg) in Patients With Moderate to Severe COPD Using Salbutamol (200 μg) and Salmeterol/Fluticasone (50/500 μg) as Active Controls
Brief Title: Study to Determine the Onset of Action of Indacaterol in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CQAB149B2307; EUDRACT: 2007-006189-14
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; indacaterol; adults
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Salmeterol Xinafoate; Fluticasone; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ind 150μg, Salm/flut, Ind 300μg, Placebo, Salbut (Experimental): Participants received a single dose of each treatment from Period I - V in the following order, separated by a washout period of 4-7 days: Indacaterol 150 μg (Ind 150μg), Salmeterol/fluticasone 50/500 μg (Salm/flut), Indacaterol 300 μg (Ind 300μg), Placebo, Salbutamol 200 μg (Salbut). At each treatment visit, participants received the specified treatment and 2 placebo inhalations (one inhalation from the SDDPI, and one inhalation from each of the two MDDPIs) to maintain blinding. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol/fluticasone (50/500 μg); Drug: Salbutamol (200 µg); Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol/fluticasone; Drug: Placebo to salbutamol
- Ind 300μg, Ind 150μg, Salbut, Salm/flut, Placebo (Experimental): Participants received a single dose of each treatment from Period I - V in the following order, separated by a washout period of 4-7 days: Indacaterol 300 μg (Ind 300μg), Indacaterol 150 μg (Ind 150μg), Salbutamol 200 μg (Salbut), Salmeterol/fluticasone 50/500 μg (Salm/flut), Placebo. At each treatment visit, participants received the specified treatment and 2 placebo inhalations (one inhalation from the SDDPI, and one inhalation from each of the two MDDPIs) to maintain blinding. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol/fluticasone (50/500 μg); Drug: Salbutamol (200 µg); Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol/fluticasone; Drug: Placebo to salbutamol
- Salm/flut, Placebo, Ind 150μg, Salbut, Ind 300μg (Experimental): Participants received a single dose of each treatment from Period I - V in the following order, separated by a washout period of 4-7 days: Salmeterol/fluticasone 50/500 μg (Salm/flut), Placebo, Indacaterol 150 μg (Ind 150μg), Salbutamol 200 μg (Salbut), Indacaterol 300 μg (Ind 300μg). At each treatment visit, participants received the specified treatment and 2 placebo inhalations (one inhalation from the SDDPI, and one inhalation from each of the two MDDPIs) to maintain blinding. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol/fluticasone (50/500 μg); Drug: Salbutamol (200 µg); Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol/fluticasone; Drug: Placebo to salbutamol
- Salbut, Ind 300μg, Placebo, Ind 150μg, Salm/flut (Experimental): Participants received a single dose of each treatment from Period I - V in the following order, separated by a washout period of 4-7 days: Salbutamol 200 μg (Salbut), Indacaterol 300 μg (Ind 300μg), Placebo, Indacaterol 150 μg (Ind 150μg), Salmeterol/fluticasone 50/500 μg (Salm/flut). At each treatment visit, participants received the specified treatment and 2 placebo inhalations (one inhalation from the SDDPI, and one inhalation from each of the two MDDPIs) to maintain blinding. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol/fluticasone (50/500 μg); Drug: Salbutamol (200 µg); Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol/fluticasone; Drug: Placebo to salbutamol
- Placebo, Salbut, Salm/flut , Ind 300μg, Ind 150μg (Experimental): Participants received a single dose of each treatment from Period I - V in the following order, separated by a washout period of 4-7 days: Placebo, Salbutamol 200 μg (Salbut), Salmeterol/fluticasone 50/500 μg (Salm/flut), Indacaterol 300 μg (Ind 300μg), Indacaterol 150 μg (Ind 150μg). At each treatment visit, participants received the specified treatment and 2 placebo inhalations (one inhalation from the SDDPI, and one inhalation from each of the two MDDPIs) to maintain blinding. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
  Interventions: Drug: Indacaterol; Drug: Salmeterol/fluticasone (50/500 μg); Drug: Salbutamol (200 µg); Drug: Placebo to Indacaterol; Drug: Placebo to Salmeterol/fluticasone; Drug: Placebo to salbutamol

INTERVENTIONS:
Drug: Indacaterol — Indacaterol 150 and 300 μg, delivered via single-dose dry-powder inhaler (SDDPI)
  Other Names: Arcapta; Neohaler
Drug: Salmeterol/fluticasone (50/500 μg) — Salmeterol/fluticasone 50/500 μg fixed-dose combination delivered via manufacturer's proprietary Multi-Dose Dry-Powder Inhaler (MDDPI).
Drug: Salbutamol (200 µg) — Salbutamol 200 μg delivered via manufacturer's proprietary Multi-Dose Dry-Powder Inhaler (MDDPI).
Drug: Placebo to Indacaterol — Placebo to indacaterol delivered via SDDPI
Drug: Placebo to Salmeterol/fluticasone — Placebo to salmeterol/fluticasone delivered via MDDPI
Drug: Placebo to salbutamol — Placebo to salbutamol delivered via MDDPI

SUMMARY:
This study will evaluate the onset of action of indacaterol (150 and 300 µg) as compared to placebo, salbutamol 200 µg and salmeterol/fluticasone 50/500 µg

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥40 years, who have signed an Informed Consent Form prior to initiation of any study-related procedure
* Patients with a diagnosis of Chronic Obstructive Pulmonary Disease (COPD) (moderate-to-severe as classified by the GOLD Guidelines, 2006) and:

  * Smoking history of at least 20 pack years
  * Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) <80% and ≥30% of the predicted normal value.
  * Post-bronchodilator FEV1/Forced Vital Capacity (FVC) < 70%, where FVC is forced vital capacity ('Post-' refers to 15-30 minutes after inhalation of 400 μg of salbutamol at Visit 2)

Exclusion Criteria:

* Pregnant / nursing women or women of child-bearing potential
* Long term oxygen therapy (more than 15 hours per day) on a daily basis for chronic hypoxemia
* Patients hospitalized for COPD exacerbation in 6 weeks prior to Visit 2 and up to Visit 3
* Respiratory tract infection within 6 weeks prior to Visit 2 and up to Visit 3
* Concomitant pulmonary disease, pulmonary tuberculosis (unless chest x-ray confirms no longer active) or clinically significant bronchiectasis
* Any history of asthma, including: blood eosinophil count >400/mm3; onset of asthma symptoms prior to age 40 years
* History of long QT syndrome or whose QTc (Bazett's) measured at Visit 2 or Visit 3 is prolonged (>450ms for males or >470ms for females)
* Clinically relevant lab abnormalities / conditions such as (but not limited to) unstable ischemic heart disease, arrhythmia (excluding stable AF), uncontrolled hypertension, uncontrolled hypo- and hyperthyroidism, hypokalemia, hyperadrenergic state or any condition which in the investigator's opinion might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study
* Uncontrolled Type I / Type II Diabetes or blood glucose outside normal or HbA1c >8.0% of total hemoglobin measured at Visit 2
* Any patient with lung cancer or any active cancer or a history of cancer with less than 5 years disease-free survival time
* History of hypersensitivity to any of the study drugs
* Irregular day/night, waking/sleeping cycles e.g. shift workers
* Live attenuated vaccinations within 30 days prior to Visit 2
* Investigational drug within 30 days prior to Visit 2
* Known history of non-compliance or not able to use devices or perform spirometry

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (5):
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigator Site, Lafayette, Louisiana
  - Novartis Investigative Site, Saint Charles, Missouri
  - Novartis Investigative site, Shelby, North Carolina
  - Novartis Investigative Site, Beaver, Pennsylvania
- Novartis Investigative Site, Antwerp, Belgium
- Germany (8):
  - Novartis Investigative Site, Berlin
  - Novartis Investigator Site, Borstel
  - Novartis Investigative site, Dortmund
  - Novartis Investigative site, Hamburg
  - Novartis Investigative site, Hanover
  - Novartis Investigative site, Mainz
  - Novartis Investigator Site, Potsdam
  - Novartis Investigative site, Wiesbaden
- Hungary (3):
  - Novartis Investigative site, Debrecen
  - Novartis Investigative site, Deszk
  - Novartis Investigative Site, Nyíregyháza

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Ind 150μg, Salm/Flut, Ind 300μg, Placebo, Salbut | Ind 300μg, Ind 150μg, Salbut, Salm/Flut, Placebo | Salm/Flut, Placebo, Ind 150μg, Salbut, Ind 300μg | Salbut, Ind 300μg, Placebo, Ind 150μg, Salm/Flut | Placebo, Salbut, Salm/Flut , Ind 300μg, Ind 150μg
Started | 18 | 17 | 18 | 18 | 18
Completed | 18 | 17 | 17 | 18 | 17
Not Completed | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1
Period: Period 2
Arm/Group | Ind 150μg, Salm/Flut, Ind 300μg, Placebo, Salbut | Ind 300μg, Ind 150μg, Salbut, Salm/Flut, Placebo | Salm/Flut, Placebo, Ind 150μg, Salbut, Ind 300μg | Salbut, Ind 300μg, Placebo, Ind 150μg, Salm/Flut | Placebo, Salbut, Salm/Flut , Ind 300μg, Ind 150μg
Started | 18 | 17 | 17 | 18 | 17
Completed | 18 | 17 | 17 | 18 | 17
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Ind 150μg, Salm/Flut, Ind 300μg, Placebo, Salbut | Ind 300μg, Ind 150μg, Salbut, Salm/Flut, Placebo | Salm/Flut, Placebo, Ind 150μg, Salbut, Ind 300μg | Salbut, Ind 300μg, Placebo, Ind 150μg, Salm/Flut | Placebo, Salbut, Salm/Flut , Ind 300μg, Ind 150μg
Started | 18 | 17 | 17 | 18 | 17
Completed | 17 | 17 | 17 | 18 | 17
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Ind 150μg, Salm/Flut, Ind 300μg, Placebo, Salbut | Ind 300μg, Ind 150μg, Salbut, Salm/Flut, Placebo | Salm/Flut, Placebo, Ind 150μg, Salbut, Ind 300μg | Salbut, Ind 300μg, Placebo, Ind 150μg, Salm/Flut | Placebo, Salbut, Salm/Flut , Ind 300μg, Ind 150μg
Started | 17 | 17 | 17 | 18 | 17
Completed | 17 | 17 | 17 | 18 | 17
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Ind 150μg, Salm/Flut, Ind 300μg, Placebo, Salbut | Ind 300μg, Ind 150μg, Salbut, Salm/Flut, Placebo | Salm/Flut, Placebo, Ind 150μg, Salbut, Ind 300μg | Salbut, Ind 300μg, Placebo, Ind 150μg, Salm/Flut | Placebo, Salbut, Salm/Flut , Ind 300μg, Ind 150μg
Started | 17 | 17 | 17 | 18 | 17
Completed | 17 | 17 | 17 | 18 | 17
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Population: Participants were randomized to one of five treatment sequences. Each treatment sequence comprised 5 double-blind, single dose treatment periods (Periods I to V), separated by a washout period of 4-7 days. Participants received each of the 5 blinded-treatments: indacaterol 150 μg, indacaterol 300 μg, salmeterol/fluticasone 50/500 μg, salbutamol 200 μg and placebo.
Arm/Group | Total Population
Number analyzed (Participants) | 89
Age Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) at 5 Minutes Post-dose
Description: FEV1 was measured at 5 minutes after dosing with spirometry conducted according to internationally accepted standards. The time of dosing was defined as the time corresponding to the use of the first inhaler device. The primary variable was analyzed using a mixed model containing the period baseline FEV1 as covariate. The period baseline FEV1 was the average of the FEV1 value measured in the clinic at 50 and 15 min prior to the study drug administration in that period.
Time Frame: Five Minutes Post Dose
Population: Modified Intent-to-Treat (mITT) population: including all randomized patients who received at least one dose of study drug. If any of the values used in the period baseline FEV1 and FEV1 at 5 min post-dose were collected within 6 hours of rescue medication, then the individual FEV1 value was set to missing.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Indacaterol 150 µg: Participants received a single dose of Indacaterol 150 µg delivered via a Single-Dose Dry-Powder Inhaler (SDDPI), placebo to salmeterol/fluticasone delivered via Multi-Dose Dry-Powder Inhaler (MDDPI) and placebo to salbutamol delivered via MDDPI. Each treatment period lasted up to 2 hours following study drug administration and was separated from the previous treatment by a washout period of 4 to 7 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol 300 µg: Participants received a single dose of Indacaterol 300 µg delivered via a Single-Dose Dry-Powder Inhaler (SDDPI), a placebo to salmeterol/fluticasone delivered via Multi-Dose Dry-Powder Inhaler (MDDPI) and a placebo to salbutamol delivered via MDDPI. Each treatment period lasted up to 2 hours following study drug administration and was separated from the previous treatment by a washout period of 4 to 7 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Placebo: Participants received placebo to indacaterol delivered via Single-Dose Dry-Powder Inhaler (SDDPI), a placebo to salmeterol/fluticasone delivered via Multi-Dose Dry-Powder (MDDPI) and placebo to salbutamol delivered via MDDPI. Each treatment period lasted up to 2 hours following study drug administration and was separated from the previous one by a washout period of 4 to 7 days. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Salmeterol/Fluticasone: Participants received a single dose of Salmeterol/fluticasone 50/500 µg delivered via MDDPI, a placebo to indacaterol delivered via SDDPI and placebo to salbutamol delivered via MDDPI. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Salbutamol: Participants received a single dose of Salbutamol 200 µg delivered via MDDPI, a placebo to indacaterol delivered via SDDPI and placebo to salmeterol/fluticasone delivered via MDDPI. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Placebo | Salmeterol/Fluticasone | Salbutamol
Number analyzed (Participants) | 85 | 87 | 88 | 88 | 86
Liters | 1.48 (0.014) | 1.50 (0.014) | 1.38 (0.014) | 1.43 (0.014) | 1.47 (0.014)

ADVERSE EVENTS:
Time Frame: 54 days
Description: Safety population including all patients who received at least one dose of study drug.
Groups:
- Indacaterol 150 µg: Participants received a single dose of Indacaterol 150 µg delivered via a Single-Dose Dry-Powder Inhaler (SDDPI), placebo to salmeterol/fluticasone delivered via Multi-Dose Dry-Powder Inhaler (MDDPI) and placebo to salbutamol delivered via MDDPI. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Indacaterol 300 µg: Participants received a single dose of Indacaterol 300 µg delivered via Single-Dose Dry-Powder Inhaler (SDDPI), a placebo to salmeterol/fluticasone delivered via Multi-Dose Dry-Powder Inhaler (MDDPI) and placebo to salbutamol delivered via MDDPI. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
- Placebo: Participants received placebo to indacaterol delivered via SDDPI, a placebo to salmeterol/fluticasone delivered via MDDPI and placebo to salbutamol delivered via MDDPI. Daily inhaled corticosteroid treatment (if applicable) was to remain stable throughout the study. The short-acting β2-agonist salbutamol/albuterol was available for rescue use throughout the study.
Arm/Group | Indacaterol 150 µg | Indacaterol 300 µg | Salbutamol | Salmeterol/Fluticasone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/87 | 0/86 | 0/88 | 0/87
Other Adverse Events (participants affected / at risk) | 0/86 | 0/87 | 0/86 | 0/88 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.